CLINICAL TRIAL: NCT02765360
Title: Changes in Lung Ventilation With Different Modes of Non-invasive Ventilation in COPD and OHS Patients
Brief Title: EIT Study With COPD and OHS Patients (EIT Step 2)
Acronym: EIT & NIV Step
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: B&D Electromedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 187764 15/LO/1921
Record Dates: First submitted 2016-02-12; First posted 2016-05-06 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: OHS; COPD
Keywords: EIT; NIV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Each patient will be assigned to Continuous Positive Airway Pressure (CPAP), Pressure Support Ventilation (PSV) and Pressure Control Ventilation (PCV) modes in a random order with a 10 minute washout period modes.
  Interventions: Other: Treatment Group

INTERVENTIONS:
Other: Treatment Group — Participants will be established on the randomised mode of ventilation and will have continuous assessment of the following during the assessment period:
  * Electrical impedance tomography
  * EMGpara
  * SpO2
  * tcCO2
  * Pneumotachography
  * End-tidal CO2 monitoring

SUMMARY:
Patients with severe respiratory diseases such as chronic obstructive pulmonary disease (COPD) or obesity-hypoventilation syndrome (OHS) can benefit from having non-invasive ventilation (NIV). NIV consists of a machine (ventilator) that is blowing air inside a patient's airway through a mask. NIV provides patients with a bigger breath. Bigger breaths help patients to have a more oxygen and less waste gas (or carbon dioxide) in their body.

These changes can improve outcomes and quality of life. In order to provide appropriate ventilation for each patient, the ventilator can generate different types of blowing:

* Continuous positive airway pressure (CPAP) which delivers a constant flow of air through the mask
* Pressure support ventilation (PSV) which delivers a constant flow of air through the mask and, on top of that, delivers more flow when the patient begins to inhale
* Volume targeted ventilation which delivers a flow of air through the mask that is adjusted breath by breath in order to achieve a preset volume.

These different type of blowing have consequences on patient comfort as well as on the improvement of their ventilation.

To assess the improvement of the ventilation, currently blood tests are used, however, these reflect overall output and may miss more subtle changes in breathing that could affect how patients feel.

Electrical impedance tomography (EIT) is a new technology that involves wearing a belt of sensors around the chest that provides information on how well the lungs are being filled with air by the ventilator. It allows a non-invasive assessment of the effect of NIV on lung ventilation in real-time.

The investigators hope to use the EIT technology to assess in real-time patients lung ventilation when they are using the NIV. The investigators hope that EIT will provide information on which type of blowing is more effective and more comfortable than the others.

DETAILED DESCRIPTION:
Chronic lung disease can sometimes progress to the extent that patients can no longer clear the waste gas from their blood. Treatment can be offered with a mask and machine (ventilator) that helps people breathe and aims to improve their lung condition. It is common for people's lungs to be affected variably, i.e. left more than right or top of lung more than bases of lungs. The way in which the ventilator is set may affect how well the machine deals with these differences. If the lung is better ventilator patients may find the machine more comfortable and it may be more effective.

Electrical impedance tomography (EIT) is a new technology that involves wearing a belt of sensors around the chest that provides information on how well the lungs are being filled with air by the ventilator. It allows the assessment of these differences, which previously required the use of invasive equipment to obtain.

Optimising ventilator settings in the administration of non-invasive ventilation (NIV) can be improved with the addition of individual physiological data. This approach is limited due to the invasive techniques required to obtain this information, often leading to less ideal NIV settings promoting patient-ventilator asynchrony. It has been recently demonstrated by our group that all patients established on domiciliary NIV have a degree of patient-ventilator asynchrony and that the commonest type of asynchrony are triggering issues. Triggering asynchrony is promoted by mismatch between a patient's intrinsic positive end-expiratory pressure (iPEEP) and applied expiratory positive airway pressure (EPAP) with these ineffective efforts contributing to an increased work of breathing and patient discomfort. Previous strategies used to optimise patient triggering have involved the placement of oesophageal catheters in order to measure neural respiratory drive (NRD) to the diaphragm by electromyography (EMG) but again this process is invasive and often poorly tolerated. Electrical Impedance Tomography (EIT) is a non-invasive, bedside monitoring technique that provides semi-continuous, real-time information about the regional distribution of the changes in electrical resistivity of the lung tissue due to variations in ventilation in relation to a reference state.

Information is gained by repeatedly injecting small alternating electric currents (usually 5 mA) at high frequency of 50 - 80 kHz through a system of skin electrodes (usually 16) applied circumferentially around the thorax in a single plane between the 4th and 6th intercostal space. While an adjacent pair of electrodes 'injects' the current ('adjacent drive configuration'), all the remaining adjacent passive electrode pairs measure the differences in electric potential. A resistivity (impedance) image is reconstructed from this data by a mathematical algorithm using a two dimensional model and a simplified shape to represent the thoracic cross-section.

The resulting image possesses a high temporal and functional resolution making it possible to monitor dynamic physiological phenomena (e.g. delay in regional inflation or recruitment) on a breath by breath basis. It is important to realize that the EIT images are based on image reconstruction techniques that require at least one measurement on a well-defined reference state. All quantitative data are related to this reference and can only indirectly quantify (relative) changes in local lung impedance (but not absolute).

EIT can be used in mechanically ventilated patients to assess recruitment and to optimise ventilator settings to reduce risk of iatrogenic ventilator associated lung injury.

In the supine posture obese patients can generate significant levels of iPEEP that contribute to increased levels of neural respiratory drive compared with the upright posture. There has been much debate regarding the optimal ventilator strategy in patients with obesity related respiratory failure, with uncontrolled trial data to support simple continuous positive airway pressure, pressure support (PSV) NIV and volume targeted (VT) NIV. There has been no robust evidence to suggest superiority of a single mode but post hoc data suggests superior control of sleep disordered breathing in patients in pressure controlled mode. It is unclear whether the extended inspiratory time of pressure controlled mode is allowing superior gas exchange by maintaining airway distension and preventing regional collapse.

In COPD, patients' response to treatment can be influenced by disease heterogeneity with some patients showing even distribution of lung damage and others marked differences throughout the lungs. This variation can lead to significant differences in the lung mechanics in different regions with optimal NIV settings for some regions having potentially deleterious effects on neighbouring zones. It has been shown that control of hypoventilation and improved blood gas exchange is essential in order to improve outcomes with NIV in COPD but is less clear if pressure control ventilation as advocated by Windisch and colleagues is required in order to achieve this effect. Inappropriate settings of NIV can also lead to dynamic distension that results in a decrease of tidal volume and an increase in patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* On domiciliary NIV for at least 3 months
* Domiciliary NIV set up following an arterial puncture showing a PaCO2 > 6 kPa
* Compliance of > 4 hours per night
* FEV1 / FVC < 70% and FEV1 < 70% for COPD participants
* FEV1 > 70% for OHS participants
* Previous chest computed tomography for COPD participants
* BMI >35 kg/m2 for OHS participants

Exclusion Criteria:

* Pregnancy
* Aged <18, >80
* Significant physical or psychiatric comorbidity that would prevent compliance with trial protocol
* Decompensated respiratory failure (pH < 7.35)
* BMI > 50kg/m2

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Characteristics seen during ventilation in different modes of ventilation | 1 day
  What happens to the lung when ventilation on different modes

SECONDARY OUTCOMES:
Lung volumes on EIT compared with pneumotachography assessed lung volumes | 1 day
  Comparing lung volumes comparison whilst on EIT and pneumotachography
Patient ventilator asynchrony | 1 day
Neural respiratory drive (EMGpara) | 1 day
Subjective patient comfort (Visual analogue scale - VAS - Borg scale) | 1 day
Patient comfort and lung homogeneity | 1 day
  Assessment of patient comfort during ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hart, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No